CLINICAL TRIAL: NCT02450370
Title: Comparison of Symptom Response Following a Conventional Irritable Bowel Syndrome Dietary Advice Versus Low FODMAP Diet in Hong Kong Chinese Irritable Bowel Syndrome Patients
Brief Title: Diets in Symptom Relief and the Influence of Quality of Life in People With Irritable Bowel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong Sanatorium & Hospital (Industry)
Collaborators: The Hong Kong Society of Gastrointestinal Motility (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC-201405
Record Dates: First submitted 2015-05-19; First posted 2015-05-21 (Estimated); Last update posted 2018-06-25 (Actual); Status verified 2018-06

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — FODMAP Diet

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional IBS diet group (Active Comparator): Subjects in this group will follow a conventional diet for up to 10 weeks. They will receive 3 dietetic consultations at week 0,6 and 10. This diet will focus on small frequent meals, no skipping meals and dietary adjustments for bloatedness, diarrhea and constipation. Advice on intake of caffeine and alcohol will also be given. Dietary leaflets will be provided.
  Interventions: Behavioral: Conventional IBS diet group
- Low FODMAP diet group (Experimental): Subjects in this group will follow a low FODMAP diet for up to 10 weeks. Foods that are high in oligosaccharides, disaccharides, monosaccharides and polyols will be avoided. They will receive 3 dietetic consultations at week 0,6 and 10. Dietary leaflets, including meal samples and Yes/No food lists will be provided.
  Interventions: Behavioral: Low FODMAP diet

INTERVENTIONS:
Behavioral: Low FODMAP diet — Subjects in this group will follow a low FODMAP diet for up to 10 weeks. Foods that are high in oligosaccharides, disaccharides, monosaccharides and polyols will be avoided. They will receive 3 dietetic consultations at week 0,6 and 10. Dietary leaflets, including meal samples and Yes/No food lists will be provided.
  Arms: Low FODMAP diet group
Behavioral: Conventional IBS diet group — Subjects in this group will follow a conventional diet for up to 10 weeks. They will receive 3 dietetic consultations at week 0,6 and 10. This diet will focus on small frequent meals, no skipping meals and dietary adjustments for bloatedness, diarrhea and constipation. Advice on intake of caffeine and alcohol will also be given. Dietary leaflets will be provided.
  Arms: Conventional IBS diet group

SUMMARY:
Subjects with confirmed diagnosis of Irritable Bowel Syndrome will be blinded and randomly assigned to one of two groups, the low FODMAP diet or the conventional IBS diet group. They will be referred to do three hydrogen breath tests prior to diet education. Upon completion, subjects will attend dietitian consultations at Week 0, 6 and 10 for diet assessment, education and reinforcement. At Week 4 and 8, dietitians will telephone patients to check on diet compliance and answer any diet question. Two sets of questionnaires, the IBS Global Improvement Scale and the IBSQOL will be given to patients to complete before each dietitian visit at week 0, 6 and 10. Two sample t-test and Chi square test will be used to test the difference between the two groups and the association between breath tests results and responds to the two diets.

DETAILED DESCRIPTION:
1. Subjects who are interested will be interviewed and screened for IBS with Rome Ⅲ criteria by the principle investigator. Research information will be explained in length and consent form will be signed if they agreed to participate
2. Subjects will be blinded and randomly assigned to Conventional IBS diet group (A) or Low FODMAP diet group (B)
3. 3 Breath tests (lactulose, fructose, lactose) will be carried out for all subjects before diet education
4. Subjects will be asked to come to the dietitians clinic and receive the first one hour diet education (including diet assessment & diet education) and two times thirty minutes follow-up appointments with the dietitians at Week 0, 6 and 10, respectively
5. Subjects will be asked to record their food intake and signs and symptoms onto a food record book
6. Subjects will be asked to fill out the IBS Global Improvement Scale and the IBSQOL questionnaire at Week 0, 6 & 10
7. At week 4 and week 8, telephone interviews will be conducted by the dietitians to reinforce diets and answer diet questions
8. Results of IBS Global Improvement Scale and IBSQOL questionnaire will be analyzed using two sample t-test to test the difference between control and treatment group
9. Chi square test will be used to look at the association between breath tests results and responds to the two diets

ELIGIBILITY:
Inclusion Criteria:

* Adults >18 years
* Confirmed IBS (after meeting Rome Ⅲ criteria)
* Hong Kong Chinese

Exclusion Criteria:

* Age <18 years
* Pregnancy
* Other ethnicities besides Hong Kong Chinese
* Significant GI co-morbidities such as Inflammatory Bowel Disease, Coeliac disease, significant diverticular disease, history of GI cancer, GI resection and GI reconstruction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2015-05; Primary Completion 2017-11-20 (Actual); Study Completion 2017-11-20 (Actual)

PRIMARY OUTCOMES:
Improvement in IBS symptoms after adopting the low FOMDAP diet versus conventional IBS diet using IBS Global Improvement Scale | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Chow, MSc, Principal Investigator — Hong Kong Sanatorium & Hospital
Locations (1):
- Dietetic Service, HKSH, Hong Kong, Hong Kong